CLINICAL TRIAL: NCT04247152
Title: Comparison of Pre-operative Measurements With Intraoperative Aberrometry in Predicting Needed Correction for Low Toric Lens Correction in Cataract Surgery
Brief Title: Comparison of Pre-operative Measurements With Intraoperative Aberrometry in Predicting Correction for Low Toric Lens Correction in Cataract Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Research Insight LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1909 ORA vs Biometry
Record Dates: First submitted 2020-01-24; First posted 2020-01-29 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-01

CONDITIONS: Cataract Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intraoperative Aberrometry vs Preoperative Biometry (Other): Retrospective view of existing chart data.
  Interventions: Other: Intraoperative Aberrometry vs preoperative biometry

INTERVENTIONS:
Other: Intraoperative Aberrometry vs preoperative biometry — Hypothesis: Intraoperative aberrometry measures lower levels of astigmatism more accurately than preoperative biometry in patients undergoing cataract surgery.

SUMMARY:
Examination of the accuracy of toric predictive power in patients with 1.5 diopters of astigmatism or less.

DETAILED DESCRIPTION:
Based on preoperative keratometry and using the Baylor Nomogram and a standard factor for surgically-induced astigmatism, the investigators will calculate "keratometry-based total astigmatism" for each patient. This will be compared to "aberrometry-based total astigmatism", i.e. the total astigmatism measured by ORA in each case. With this information the investigators will determine in what portion of patients keratometry-based total astigmatism vs aberrometry-based total astigmatism predicts a need for astigmatism correction, (i.e., total astigmatism is greater than or equal to 0.5 D) during cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent conventional (non-femtosecond) cataract surgery and whose "data to be collected" are accessible and available from the ORA database.
* Patients whose medical records show they did not exhibit any significant ocular morbidity that would be expected to influence outcome measures.

Exclusion Criteria:

* Patients with visually significant co-morbidities (corneal, retina, optic nerve disease) that could affect their visual outcome or ability to be refracted after.
* Patients with surgical complications either during or after surgery (capsule tears, iris trauma, decentered IOL, cystoid macular edema, etc.)
* Patients with previous refractive surgery.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2019-07-22 (Actual); Primary Completion 2019-09-25 (Actual); Study Completion 2019-09-25 (Actual)

PRIMARY OUTCOMES:
Proportion of Patients requiring Astigmatism Correction | up to 3 months
  Proportion of patients requiring astigmatism correction, i.e., having need for astigmatism correction of greater than or equal to 0.5 D during cataract surgery, when measured by preoperative keratometry vs intraoperative aberrometry.

SECONDARY OUTCOMES:
Patients with Postoperative residual astigmatism 0.5 to 1.0 diopter | up to 3 months
  Looking at patients whose ORA-based total astigmatism was greater than or equal to 0.5 and less than or equal to 1.0 diopter, did patients receiving astigmatism correction have less postoperative residual astigmatism than those who did not receive astigmatism correction?
Patients with Postoperative residual astigmatism 1.0 to 1.5 diopter | up to 3 months
  Looking at patients whose ORA-based total astigmatism was greater than 1.0 and less than or equal to 1.5 diopter,m did patients receiving astigmatism correction have less postoperative residual astigmatism than those who did not receive astigmatism correction?

CONTACTS AND LOCATIONS:
Locations (1):
- Harvard Eye Associates, Laguna Hills, California, United States

IPD SHARING:
Plan to Share IPD: No